CLINICAL TRIAL: NCT04104945
Title: Volume and Dose De-Intensified Radiotherapy for p16+ Squamous Cell Carcinoma of the Oropharynx: A Multi-Centre, Single Arm Prospective Cohort Study
Brief Title: p16+ Oropharyngeal Cancer Radiation Optimization Trial Reducing Elective Treatment Volumes (PROTEcT)
Acronym: PROTEcT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Tom Baker Cancer Centre (Other); Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTEcT
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- De-intensified chemoradiotherapy (Experimental): Radiotherapy to a dose of 60 Gy to the primary tumour and involved lymph nodes and 54 Gy to subclinical regions at risk in 30 fractions. Reduced volume of elective nodal radiation.
  Interventions: Radiation: De-intensified chemoradiotherapy

INTERVENTIONS:
Radiation: De-intensified chemoradiotherapy — Radiotherapy to a dose of 60 Gy to the primary tumour and involved lymph nodes and 54 Gy to subclinical regions at risk in 30 fractions. Reduced volume of elective nodal radiation.

SUMMARY:
Volume and Dose De-Intensified Radiotherapy for p16+ Squamous Cell Carcinoma of the Oropharynx: A Multi-Centre, Single Arm Prospective Cohort Study

DETAILED DESCRIPTION:
De-intensified radiotherapy to a dose of 60 Gy to the primary tumour and involved lymph nodes and 54 Gy to subclinical regions at risk in 30 fractions. Omission of level IB lymph node regions from the elective nodal volumes.

Chemotherapy will be administered as per standard of care, consisting of concurrent cisplatin (high-dose: 100mg/m2 IV every 3 weeks or low-dose: 40mg/m2 IV every week) or cetuximab (at the discretion of medical oncologist).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older

  * Provide informed consent
  * ECOG performance status 0-2
  * Histologically confirmed squamous cell carcinoma
  * p16-positive tumor, as determined by immunohistochemistry at local hospital
  * Primary tumor site in the oropharynx (includes tonsil, soft palate, base of tongue, walls of oropharynx)
  * Eligible for curative intent treatment.
  * Smokers and non-smokers are included
  * Tumor stage (AJCC 8th edition): T1 to T3
  * Nodal stage (AJCC 8th edition): N1 to N2
  * Adequate bone marrow function, hepatic, and renal function for chemotherapy (Hemoglobin > 80 g/L; Absolute neutrophil count >1.5x109 /L, platelets > 100 x109/L; Bilirubin < 35 umol/L; AST or ALT < 3 x the upper limit of normal; serum creatinine < 130 umol/L or creatinine clearance ≥ 50 ml/min)

Exclusion Criteria:

* - Clinical, radiologic or pathologic Ib nodal involvement (including invasion into submandibular gland)
* Primary cancer with extension and involvement of the oral cavity
* Metastatic disease
* Contraindications to radiotherapy or chemotherapy
* Prior history of head and neck cancer within 5 years
* Prior head and neck radiation at any time
* Inability to attend full course of radiotherapy or follow-up visits
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2028-10-21 (Estimated); Study Completion 2028-10-21 (Estimated)

PRIMARY OUTCOMES:
Xerostomia-related quality of life | 12 months
  Measured by the Xerostomia Questionnaire (XQ), which is an 8 item self-reported xerostomia specific questionnaire. Patients rate each item on an 11 point ordinal Likert scale from 0 to 10, with higher scores indicating greater dryness or discomfort due to dryness. Item scores are added and the sum is transformed linearly to a final summary score ranging between 0 and 100, with higher scores representing greater levels of xerostomia. Based on existing literature, the mean XQ score for patients treated with standard dose and volume radiotherapy is estimated to be 52 (null hypothesis). To detect a clinically meaningful reduction of 11 points in patients treated with volume and dose de-intensified radiotherapy, with a resulting mean XQ score of 41 (alternative hypothesis), with an alpha of 0.05 and 80% power using a one-sided Wilcoxon test assuming normal distribution, 28 patients are required. Accounting for 10% dropout a total sample size of 32 patients is required.
Toxicity Criteria for Adverse Events | Baseline to 5 years
  Measured by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

OTHER OUTCOMES:
Overall survival | Baseline to 5 years
  Time from treatment initiation to death from any cause
Progression-free survival | Baseline to 5 years
  Time from treatment initiation to disease progression or death from any cause
Local, regional, and distant failure rates | Baseline to 5 years
  Time from treatment initiation to local, regional, and distant failure
Swallowing function | 12 months
  Measured by fibre-optic endoscopic evaluation of swallowing (FEES) or modified barium swallow (MBS)
#1 Quality of life | Baseline to 5 years
  The primary study endpoint is the Xerostomia Questionnaire (XQ), an 8 item self-reported xerostomia specific questionnaire. Patients rate each item on an 11 point ordinal Likert scale from 0 to 10, with higher scores indicating greater dryness or discomfort due to dryness. Item scores are added and the sum is transformed linearly to a final summary score ranging between 0 and 100, with higher scores representing greater levels of xerostomia.
#2 Quality of life | Baseline to 5 years
  Measured by the MD Anderson Symptom Inventory - Head & Neck (MDASI-HN); a questionnaire used to assess the severity of head and neck cancer-related symptoms and their impact on six daily activities (general activity, mood, work, relations with others, walking, and enjoyment of life). Severity of symptoms are assessed on a 0-10 numerical scale, with 0 being "not present" and 10 being "as bad as you can imagine." The ratings can be averaged into several subscale scores: mean core symptom severity (13 core symptom items), mean module symptom severity (additional module symptom items if using a module), mean total symptom severity (13 core symptom items plus additional module symptom items if using a module), and mean interference (6 interference items only). The interference with daily activities is rated on a 0-10 numerical scale, 0 being "did not interfere" and 10 being "interfered completely." The mean of the interference items can be used to represent overall symptom distress.
#3 Quality of life | Baseline to 5 years
  Measured by the MD Anderson Dysphagia Inventory (MDADI), which is a 20 item self-administered questionnaire designed for evaluating the impact of dysphagia on the QOL of patients with head and neck cancer. Five responses (strongly agree, agree, no opinion, disagree, and strongly disagree) are available to each question and are scored on a scale of 1 to 5. The MDADI quantifies an individual's global (G), physical (P), emotional (E), and functional (F) perceptions of their swallowing ability. Two summary scores can be obtained: 1) global and 2) composite. The global scale is a single question, which is scored individually to assess the overall impact that swallowing abilities have on QOL. The composite MDADI score summarizes overall performance on remaining 19 items of the MDADI, as a weighted average of the P, E, and F subscales. MDADI scores are normalized to range from 20 (extremely low functioning) to 100 (high functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Quon, MD, Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No